CLINICAL TRIAL: NCT01539291
Title: A Phase 3, Double-Blind Extension Study Evaluating the Efficacy and Safety of Two Different Dose Levels of Single-Agent Idelalisib (GS-1101) for Previously Treated Chronic Lymphocytic Leukemia A Companion Trial to Study GS-US-312-0116: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy and Safety of Idelalisib (GS-1101) in Combination With Rituximab for Previously Treated Chronic Lymphocytic Leukemia
Brief Title: Extension Study of Idelalisib in Participants With Chronic Lymphocytic Leukemia (CLL) Who Participated in GS-US-312-0116 (NCT01539512)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-312-0117; 2011-006293-72 (EudraCT Number)
Record Dates: First submitted 2012-02-12; First posted 2012-02-27 (Estimated); Results first posted 2019-08-20 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: CLL; CAL-101; CAL 101; GS-1101; GS 1101; PI3K; Leukemia; GS-US-312-0116; idelalisib
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia | interventions — idelalisib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- High-dose Idelalisib (Experimental): Participants will receive idelalisib 300 mg twice daily (600 mg per day).
  Interventions: Drug: Idelalisib
- Standard-dose Idelalisib (Experimental): Participants will receive idelalisib 150 mg twice daily (300 mg per day)
  Interventions: Drug: Idelalisib

INTERVENTIONS:
Drug: Idelalisib — Idelalisib tablet(s) administered orally twice daily
  Other Names: Zydelig®; GS-1101; CAL 101

SUMMARY:
The primary objective of this extension study (GS-US-312-0117) that is a companion study to Study GS-US-312-0116 (NCT01539512), is to evaluate the effect of idelalisib on the onset, magnitude, and duration of tumor control. Randomization was done in study GS-US-312-0116, and carried forward to study GS-US-312-117.

ELIGIBILITY:
Key Inclusion Criteria:

* Individuals in the primary Phase 3 study (Study GS-US-312-0116) who are compliant
* Tolerating primary study therapy

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2012-10-03 (Actual); Primary Completion 2018-05-21 (Actual); Study Completion 2018-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (45):
- United States (30):
  - Clearview Cancer Institute, Huntsville, Alabama
  - Arizona Oncology Associates, Tucson, Arizona
  - University of California, San Diego - Moores Cancer Center, La Jolla, California
  - Ventura County Hematology Oncology Specialists, Oxnard, California
  - UCLA, Santa Monica, California
  - Stanford Cancer Center, Stanford, California
  - Rocky Mountain Blood and Marrow Transplant Program, Denver, Colorado
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Georgetown University Medical Center Lombardi Cancer Center, Washington D.C., District of Columbia
  - Collaborative Research Group, Boynton Beach, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Northwestern University, Chicago, Illinois
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Weill Cornell Medical College, New York, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Willamette Valley Cancer Center, Springfield, Oregon
  - Northwest Cancer Specialists, PC, Tualatin, Oregon
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology, P.A., Fort Worth, Texas
  - M.D. Anderson Cancer Center, Houston, Texas
  - Cancer Care Network of South Texas, San Antonio, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc., Roanoke, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Yakima Valley Memorial Hospital/North Star Lodge, Yakima, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- France (2):
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Henri Becquerel, Rouen
- Germany (2):
  - Universitätsklinikum Köln, Cologne
  - Hämatologische und Internistische Gemeinschaftspraxis Dres. Eckart / Häcker, Erlangen
- Italy (2):
  - Ospedale San Raffaele S.r.l., Milan
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Torino
- United Kingdom (9):
  - Royal Bournemouth Hospital, Bournemouth
  - Addenbrooke's Hospital, Cambridge
  - Dorset County Hospital, Dorchester
  - Northwick Park Hospital, Harrow
  - St James's University Hospital, Leeds
  - Royal Liverpool University Hospital, Liverpool
  - Hammersmith Hospital, London
  - Princess Royal University Hospital, Orpington
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Result] Coutre SE, Furman RR, Sharman, JP, Cheson BD, Pagel JM, Hillmen P, et al. Second Interim Analysis of a Phase 3 Study of Idelalisib (Zydelig®) Plus Rituximab for Relapsed Chronic Lymphocytic Leukemia: Efficacy Analysis in Patient Subpopulations with Del(17p) and Other Adverse Prognostic Factors. Blood 2014; 124 (21):330
- [Result] Sharman JP, Coutre SE, Furman RR, Cheson BD, Pagel JM, Hillmen P, et al. Efficacy of Idelalisib in CLL Subpopulations Harboring Del(17p) and Other Adverse Prognostic Factors: Results from a Phase 3, Randomized, Double-blind, Placebo-controlled Trial [Poster 7011]. American Society of Clinical Oncology (ASCO) 50th Annual Meeting; 2014 May 30-June 3; Chicago, IL. J Clin Oncol 32:5s, 2014 (suppl; abstr 7011)
- [Result] Sharman JP, Coutre SE, Furman RR, Cheson BD, Pagel JM, Hillmen P, Barrientos JC, Zelenetz AD, Kipps TJ, Flinn IW, Ghia P, Eradat H, Ervin T, Lamanna N, Coiffier B, Pettitt AR, Ma S, Tausch E, Cramer P, Huang J, Mitra S, Hallek M, O'Brien SM, Stilgenbauer S. Final Results of a Randomized, Phase III Study of Rituximab With or Without Idelalisib Followed by Open-Label Idelalisib in Patients With Relapsed Chronic Lymphocytic Leukemia. J Clin Oncol. 2019 Jun 1;37(16):1391-1402. doi: 10.1200/JCO.18.01460. Epub 2019 Apr 17. PMID 30995176

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States and Europe. The first participant was screened on 03 October 2012. The last study visit occurred on 29 June 2018.
Pre-assignment Details: Participants must have been enrolled in Gilead-sponsored Study GS-US-312-0116 (NCT01539512) to be eligible to continued access to idelalisib (IDL) in this study.
Groups:
- IDL+R to IDL 150 mg: Participants received IDL 150 mg tablet twice daily plus rituximab (R) (8 infusions intravenously) in Study GS-US-312-0116 and may have entered Study GS-US-312-0117 to receive IDL 150 mg tablet twice daily.
- IDL+R (PD) to IDL 300 mg: Participants received IDL 150 mg tablet twice daily plus rituximab (8 infusions intravenously) in Study GS-US-312-0116 and met the primary endpoint of progressive disease (PD) and entered Study GS-US-312-0117 to receive IDL 300 mg tablet twice daily. Due to the small number of participants in this group, data from this group were combined with the IDL+R to IDL 150 mg group for Baseline Characteristics and Outcome Measures sections.
- Placebo+R (PD) to IDL 150 mg: Participants received placebo tablet twice daily plus rituximab (8 infusions intravenously) in Study GS-US-312-0116 and met the primary endpoint of PD and entered Study GS-US-312-0117 to receive IDL 150 mg tablet twice daily.
- Placebo+R to IDL 150 mg: Participants received placebo tablet twice daily plus rituximab (8 infusions intravenously) in Study GS-US-312-0116 and entered Study GS-US-312-0117 to receive IDL 150 mg tablet twice daily.
Period: Study GS-US-312-0116
Arm/Group | IDL+R to IDL 150 mg | IDL+R (PD) to IDL 300 mg | Placebo+R (PD) to IDL 150 mg | Placebo+R to IDL 150 mg
Started | 106 (Started = Randomized in Study GS-US-312-0116.) | 4 (Started = Randomized in Study GS-US-312-0116.) | 42 (Started = Randomized in Study GS-US-312-0116.) | 44 (Started = Randomized in Study GS-US-312-0116.)
Completed | 81 (Completed = Met Primary Endpoint (reason as determined by investigator) or finished study period.) | 4 (Completed = Met Primary Endpoint (reason as determined by investigator) or finished study period.) | 42 (Completed = Met Primary Endpoint (reason as determined by investigator) or finished study period.) | 44 (Completed = Met Primary Endpoint (reason as determined by investigator) or finished study period.)
Not Completed | 25 | 0 | 0 | 0
Not completed — Adverse Event | 9 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 12 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 2 | 0 | 0 | 0
Not completed — Other | 1 | 0 | 0 | 0
Period: Study GS-US-312-0117
Arm/Group | IDL+R to IDL 150 mg | IDL+R (PD) to IDL 300 mg | Placebo+R (PD) to IDL 150 mg | Placebo+R to IDL 150 mg
Started | 71 (Started = Completed GS-US-312-0116 and Enrolled in GS-US-312-0117.) | 4 (Started = Completed GS-US-312-0116 and Enrolled in GS-US-312-0117.) | 42 (Started = Completed GS-US-312-0116 and Enrolled in GS-US-312-0117.) | 44 (Started = Completed GS-US-312-0116 and Enrolled in GS-US-312-0117.)
Completed | 30 (Completed = Met Primary Endpoint (reason as determined by investigator) or finished study period.) | 2 (Completed = Met Primary Endpoint (reason as determined by investigator) or finished study period.) | 20 (Completed = Met Primary Endpoint (reason as determined by investigator) or finished study period.) | 18 (Completed = Met Primary Endpoint (reason as determined by investigator) or finished study period.)
Not Completed | 41 | 2 | 22 | 26
Not completed — Adverse Event | 22 | 1 | 9 | 12
Not completed — Physician Decision | 9 | 0 | 6 | 4
Not completed — Withdrawal by Subject | 5 | 0 | 6 | 4
Not completed — Study Terminated by Sponsor | 3 | 0 | 0 | 5
Not completed — Other | 2 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set included participants in the Intent-to-Treat (ITT) Analysis Set (all participants randomized in Study GS-US-312-0116) who received ≥ 1 dose of IDL, with treatment assignments designated according to randomization in Study GS-US-312-0116. Baseline data presented were collected at the beginning of Study GS-US-312-0116.
Groups:
- IDL+R to IDL: Participants received IDL 150 mg tablet twice daily plus rituximab (8 infusions intravenously) in Study GS-US-312-0116 and may have entered Study GS-US-312-0117 to receive IDL 150 mg or 300 mg tablet twice daily. Due to the small number of participants in the IDL+R (PD) to IDL 300 mg group, data from this group were combined with the IDL+R to IDL 150 mg group for Baseline Characteristics and Outcome Measures sections.
- Total: Total of all reporting groups
Arm/Group | IDL+R to IDL | Placebo+R (PD) to IDL 150 mg | Placebo+R to IDL 150 mg | Total
Number analyzed (Participants) | 110 | 42 | 44 | 196
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 21 | 13 | 10 | 44
  ≥ 65 years | 89 | 29 | 34 | 152
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 11 | 18 | 63
  Male | 76 | 31 | 26 | 133
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 3 | 1 | 1 | 5
  Ethnicity: Not Hispanic or Latino | 101 | 39 | 42 | 182
  Ethnicity: Not Permitted | 6 | 2 | 1 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 100 | 37 | 40 | 177
  Race: Black or African American | 3 | 0 | 3 | 6
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Race: Asian | 0 | 0 | 0 | 0
  Race: American Indian or Alaska Native | 0 | 0 | 0 | 0
  Race: Other | 2 | 2 | 0 | 4
  Race: Not Permitted | 5 | 3 | 1 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 80 | 38 | 30 | 148
  United Kingdom | 18 | 3 | 6 | 27
  Italy | 2 | 1 | 4 | 7
  France | 3 | 0 | 1 | 4
  Germany | 7 | 0 | 3 | 10
17p Deletion and/or TP53 Mutation Status [Count of Participants; unit: Participants]
  Either | 46 | 21 | 14 | 81
  Neither | 64 | 21 | 30 | 115
Immunoglobulin heavy chain variable region (IgHV) Mutation Status [Count of Participants; unit: Participants]
  Mutated | 19 | 6 | 7 | 32
  Unmutated | 91 | 36 | 37 | 164
Karnofsky Performance Status (KPS) [Count of Participants; unit: Participants] — KPS is a tool used to measure the ability to perform ordinary tasks. The score ranges from 0 to 100, with a higher score indicating that the participant is better able to carry out daily activities.
  Participants
    KPS = 40 | 1 | 0 | 0 | 1
    KPS = 50 | 3 | 1 | 0 | 4
    KPS = 60 | 6 | 2 | 0 | 8
    KPS = 70 | 20 | 4 | 4 | 28
    KPS = 80 | 42 | 19 | 20 | 81
    KPS = 90 | 23 | 12 | 12 | 47
    KPS = 100 | 15 | 4 | 8 | 27

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the interval from the start of study therapy to the earlier of the first documentation of definitive disease progression or death from any cause; definitive disease progression is chronic lymphocytic leukemia (CLL) progression based on standard criteria other than lymphocytosis alone. PFS was analyzed using Kaplan-Meier (KM) estimates.
Time Frame: GS-US-312-0116 Baseline to end of study GS-US-312-0117 (maximum: up to 67.6 months)
Population: Full Analysis Set included participants in the Intent-to-Treat (ITT) Analysis Set (all participants randomized in Study GS-US-312-0116) who received ≥ 1 dose of IDL, with treatment assignments designated according to randomization in Study GS-US-312-0116.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | IDL+R to IDL | Placebo+R (PD) to IDL 150 mg | Placebo+R to IDL 150 mg
Number analyzed (Participants) | 110 | 42 | 44
months | 20.3 [17.3 to 26.3] | 6.9 [4.1 to 10.7] | 16.2 [8.8 to 26.2]

2. Primary Outcome: Safety: Percentage of Participants With Any Treatment-Emergent Adverse Events (TEAE), ≥ Grade 3 TEAE, Study Drug-Related TEAE, ≥ Grade 3 Study Drug-Related TEAE, Serious TEAE, Study Drug-Related Serious TEAE, and TEAE Leading to Study Drug Discontinuation
Description: The TEAEs were defined as events in a given study period that met one of the following criteria:
  * Events with onset dates on or after the start of treatment and up to 30 days after the permanent discontinuation of the study treatment.
  * The continuing adverse events (AEs) diagnosed prior to the start of treatment and worsened in severity grade, or non-serious AEs at baseline which became serious, or AEs resulting in treatment discontinuation after the start of treatment.
  The severity of AEs was graded by the investigator according to the common terminology criteria for adverse events (CTCAE), Version 4.03, whenever possible. The relationship of an AE to study drug (idelalisib) was assessed using clinical judgment by the investigator, describing the event as either unrelated or related. Events for which the investigator did not record relationship to study drug were considered related to study drug.
Time Frame: First IDL dose date in study GS-US-312-0116 or GS-US-312-0117 to last IDL dose date in study GS-US-312-0117 (maximum: 67.3 months) plus 4 weeks
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | IDL+R to IDL | Placebo+R (PD) to IDL 150 mg | Placebo+R to IDL 150 mg
Number analyzed (Participants) | 110 | 42 | 44
percentage of participants
  Any TEAE | 98.2 | 100.0 | 97.7
  ≥ Grade 3 TEAE | 90.9 | 88.1 | 90.9
  Study Drug-Related TEAE | 68.2 | 59.5 | 72.7
  ≥ Grade 3 Study Drug-Related TEAE | 47.3 | 45.2 | 45.5
  Serious TEAE | 80.9 | 81.0 | 72.7
  Study Drug-Related Serious TEAE | 35.5 | 26.2 | 29.5
  TEAE Leading to Study Drug Discontinuation | 47.3 | 64.3 | 50.0

3. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants who achieved a complete response (CR) or partial response (PR). The determination of CLL response and progression were based on standardized International Workshop on Chronic Lymphocytic Leukemia (IWCLL) criteria, as specifically modified for this study to reflect current recommendations which considered the mechanism of action of idelalisib and similar drugs. CR and PR are defined in Protocol Amendment 9, Sections 7.5.1 and 7.5.2.
Time Frame: GS-US-312-0116 Baseline to end of study GS-US-312-0117 (maximum: up to 67.6 months)
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IDL+R to IDL | Placebo+R (PD) to IDL 150 mg | Placebo+R to IDL 150 mg
Number analyzed (Participants) | 110 | 42 | 44
percentage of participants | 85.5 [77.5 to 91.5] | 47.6 [32.0 to 63.6] | 68.2 [52.4 to 81.4]

4. Secondary Outcome: Lymph Node Response Rate
Description: Lymph node response rate was defined as the percentage of participants who achieved a ≥ 50% decrease from baseline in the sum of the products of the greatest perpendicular diameters (SPD) of index lymph nodes.
Time Frame: GS-US-312-0116 Baseline to end of study GS-US-312-0117 (maximum: up to 67.6 months)
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IDL+R to IDL | Placebo+R (PD) to IDL 150 mg | Placebo+R to IDL 150 mg
Number analyzed (Participants) | 106 | 36 | 43
percentage of participants | 97.2 [92.0 to 99.4] | 77.8 [60.8 to 89.9] | 83.7 [69.3 to 93.2]

5. Secondary Outcome: Complete Response (CR) Rate
Description: CR rate was defined as the percentage of participants who achieved a CR (full definition in Protocol Amendment 9, Section 7.5.1). The determination of CLL response and progression were based on standardized IWCLL criteria, as specifically modified for this study to reflect current recommendations which considered the mechanism of action of idelalisib and similar drugs.
Time Frame: GS-US-312-0116 Baseline to end of study GS-US-312-0117 (maximum: up to 67.6 months)
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | IDL+R to IDL | Placebo+R (PD) to IDL 150 mg | Placebo+R to IDL 150 mg
Number analyzed (Participants) | 110 | 42 | 44
percentage of participants | 0.9 | 0.0 | 0.0

6. Secondary Outcome: Time to Response (TTR)
Description: TTR was defined as the time interval from start of study therapy to the first documentation of CR or PR.
Time Frame: GS-US-312-0116 Baseline to end of study GS-US-312-0117 (maximum: up to 67.6 months)
Population: Participants in the Full Analysis Set who achieved a CR or PR were analyzed.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | IDL+R to IDL | Placebo+R (PD) to IDL 150 mg | Placebo+R to IDL 150 mg
Number analyzed (Participants) | 94 | 20 | 30
months | 2.1 [1.9 to 3.8] | 3.6 [1.9 to 4.0] | 2.8 [1.9 to 4.2]

7. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time interval from the first documentation of CR or PR to the earlier of the first documentation of definitive disease progression or death from any cause. DOR was analyzed using KM estimates.
Time Frame: From first documentation of CR or PR to end of study GS-US-312-0117 (maximum: up to 67.6 months)
Population: Participants in the Full Analysis Set who achieved a CR or PR were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | IDL+R to IDL | Placebo+R (PD) to IDL 150 mg | Placebo+R to IDL 150 mg
Number analyzed (Participants) | 94 | 20 | 30
months | 21.4 [16.6 to 26.1] | 11.0 [3.3 to NA] — NA = Too few events to estimate the upper limit of the confidence interval. | 17.6 [13.2 to 37.7]

8. Secondary Outcome: Best Percent Change in Lymph Node Area
Description: The best percent change from baseline in lymph node area (SPD) was defined as the largest decrease in tumor size during the study. The baseline SPD was the last value prior to the baseline reference date. For the participants who only had increases in tumor size from baseline, the smallest increase was considered as the best change from baseline in SPD.
Time Frame: GS-US-312-0116 Baseline to end of study GS-US-312-0117 (maximum: up to 67.6 months)
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | IDL+R to IDL | Placebo+R (PD) to IDL 150 mg | Placebo+R to IDL 150 mg
Number analyzed (Participants) | 106 | 36 | 43
percent change | -80.1 [-86.1 to -70.5] | -69.7 [-79.5 to -53.7] | -71.4 [-80.4 to -62.7]

9. Secondary Outcome: Splenomegaly Response Rate
Description: Splenomegaly response rate was defined as the percentage of participants with baseline splenomegaly who achieved an on-study normalization or a 50% decrease (minimum 2 cm) from baseline in the enlargement of the splenic longest vertical dimension (LVD) (by imaging).
Time Frame: GS-US-312-0116 Baseline to end of study GS-US-312-0117 (maximum: up to 67.6 months)
Population: Participants in the Full Analysis Set who had splenomegaly at baseline and at least 1 evaluable postbaseline spleen measurement were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IDL+R to IDL | Placebo+R (PD) to IDL 150 mg | Placebo+R to IDL 150 mg
Number analyzed (Participants) | 76 | 23 | 24
percentage of participants | 80.3 [69.5 to 88.5] | 47.8 [26.8 to 69.4] | 66.7 [44.7 to 84.4]

10. Secondary Outcome: Hepatomegaly Response Rate
Description: Hepatomegaly response rate was defined as the percentage of participants with baseline hepatomegaly who achieved an on-study normalization or a 50% decrease (minimum 2 cm) from baseline in the hepatic LVD (by imaging).
Time Frame: GS-US-312-0116 Baseline to end of study GS-US-312-0117 (maximum: up to 67.6 months)
Population: Participants in the Full Analysis Set who had hepatomegaly at baseline and at least 1 evaluable postbaseline liver measurement were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IDL+R to IDL | Placebo+R (PD) to IDL 150 mg | Placebo+R to IDL 150 mg
Number analyzed (Participants) | 54 | 22 | 20
percentage of participants | 63.0 [48.7 to 75.7] | 36.4 [17.2 to 59.3] | 30.0 [11.9 to 54.3]

11. Secondary Outcome: Absolute Lymphocyte Count (ALC) Response Rate
Description: ALC response rate was defined as the percentage of participants with baseline lymphocytosis (ALC ≥ 4 x 10^9 cells/L) who achieved an on-study ALC < 4 x 10^9 cells/L or demonstrated a ≥ 50% decrease in ALC from baseline; ALC values within 4 weeks post-baseline were excluded from the ALC response rate evaluation.
Time Frame: GS-US-312-0116 Baseline to end of study GS-US-312-0117 (maximum: up to 67.6 months)
Population: Participants in the Full Analysis Set who had lymphocytosis (ALC ≥ 4 × 10^9/L) at baseline and at least 1 evaluable postbaseline value were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IDL+R to IDL | Placebo+R (PD) to IDL 150 mg | Placebo+R to IDL 150 mg
Number analyzed (Participants) | 88 | 27 | 34
percentage of participants | 94.3 [87.2 to 98.1] | 66.7 [46.0 to 83.5] | 64.7 [46.5 to 80.3]

12. Secondary Outcome: Platelet Response Rate
Description: Platelet response rate was defined as the percentage of participants with baseline thrombocytopenia (platelet count < 100 x 10^9/L) who achieved an on-study platelet count ≥ 100 x 10^9/L or demonstrated a ≥ 50% increase in platelet count from baseline; platelet values within 4 weeks post-baseline or after 8 days post transfusion were excluded from the platelet response rate evaluation.
Time Frame: GS-US-312-0116 Baseline to end of study GS-US-312-0117 (maximum: up to 67.6 months)
Population: Participants in the Full Analysis Set who had thrombocytopenia (platelet count < 100 × 10^9/L) at baseline and at least 1 evaluable postbaseline value were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IDL+R to IDL | Placebo+R (PD) to IDL 150 mg | Placebo+R to IDL 150 mg
Number analyzed (Participants) | 50 | 23 | 10
percentage of participants | 98.0 [89.4 to 99.9] | 73.9 [51.6 to 89.8] | 100.0 [69.2 to 100.0]

13. Secondary Outcome: Hemoglobin Response Rate
Description: Hemoglobin response rate was defined as the percentage of participants with baseline anemia (hemoglobin < 110 g/L [11.0 g/dL]) who achieved an on-study hemoglobin ≥ 110 g/L (11.0 g/dL) or demonstrated a ≥ 50% increase in hemoglobin from baseline; hemoglobin values within 4 weeks post-baseline or after 4 weeks of receiving packed cell/whole blood transfusion or after 6 weeks of receiving exogenous growth factors (eg, darbepoetin alfa) were excluded from the hemoglobin response evaluation.
Time Frame: GS-US-312-0116 Baseline to end of study GS-US-312-0117 (maximum: up to 67.6 months)
Population: Participants in the Full Analysis Set who had anemia (hemoglobin < 110 g/L [11 g/dL]) at baseline and at least 1 evaluable postbaseline value were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IDL+R to IDL | Placebo+R (PD) to IDL 150 mg | Placebo+R to IDL 150 mg
Number analyzed (Participants) | 59 | 24 | 11
percentage of participants | 83.1 [71.0 to 91.6] | 45.8 [25.6 to 67.2] | 81.8 [48.2 to 97.7]

14. Secondary Outcome: Neutrophil Response Rate
Description: Neutrophil response rate was defined as the percentage of participants with baseline neutropenia (absolute neutrophil count [ANC] ≤ 1.5 x 10^9/L) who achieved an ANC > 1.5 x 10^9/L or demonstrated a ≥ 50% increase in ANC from baseline; ANC values within 4 weeks of post-baseline or after 2 weeks of receiving exogenous growth factors (eg, filgrastim, granulocyte-colony stimulating factor [G-CSF], lenograstim) or after 4 weeks of receiving Neulasta® were excluded from response evaluation.
Time Frame: GS-US-312-0116 Baseline to end of study GS-US-312-0117 (maximum: up to 67.6 months)
Population: Participants in the Full Analysis Set who had neutropenia (ANC ≤ 1.5 × 10^9/L) at baseline and at least 1 evaluable postbaseline value were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IDL+R to IDL | Placebo+R (PD) to IDL 150 mg | Placebo+R to IDL 150 mg
Number analyzed (Participants) | 27 | 11 | 6
percentage of participants | 96.3 [81.0 to 99.9] | 90.9 [58.7 to 99.8] | 100.0 [54.1 to 100.0]

15. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time interval from start of study therapy to death from any cause. Overall survival was analyzed using KM estimates. Data presented includes all available survival information from Study GS-US-312-0116 (including data in long-term follow-up) and Study GS-US-312-0117 (including any data in long-term follow-up) up to the database finalization dates. Data from surviving participants were censored at the last time that the participant was known to be alive on study or long-term follow-up. Data presented includes all participants who were randomized to Study GS-US-312-0116 regardless if they entered Study GS-US-312-0117 or not.
Time Frame: GS-US-312-0116 Baseline to end of study GS-US-312-0117 (maximum: up to 67.6 months)
Population: Per the analysis plan, overall survival data was analyzed in the ITT Analysis Set (participants who were randomized in the study) by treatment group according to the original randomization in Study GS-US-312-0116, regardless of whether participants received any study drug, or received a different regimen from the regimen they were randomized to.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- IDL+R: Participants were randomized to receive IDL 150 mg tablet twice daily plus rituximab (8 infusions intravenously) in Study GS-US-312-0116.
- Placebo+R: Participants were randomized to receive placebo tablet twice daily plus rituximab (8 infusions intravenously) in Study GS-US-312-0116.
Arm/Group | IDL+R | Placebo+R
Number analyzed (Participants) | 110 | 110
months | 40.6 [28.5 to 57.3] | 34.6 [16.0 to NA] — NA = Too few events to estimate the upper limit of the confidence interval.

16. Secondary Outcome: Best Change From Baseline in Health-Related Quality of Life (HRQL) Domain and Symptom Scores Based on the Functional Assessment of Cancer Therapy-Leukemia (FACT-Leu) Questionnaire
Description: The FACT-Leu questionnaire included subscales for physical well-being (PWB, 7 items), social/family well-being (SWB, 7 items), emotional well-being (EWB, 6 items), functional well-being (FWB, 7 items), and additional concerns or Leukemia-Specific Subscale (LeuS, 17 items). The FACT-Leu scoring guide identified those negatively stated items that must have been reversed before being added to obtain subscale totals. Negatively stated items were reversed by subtracting the response from "4". After reversing proper items, all subscale items were summed to get total subscale scores with the range of 0-28, 0-28, 0-24, 0-28, 0-68 for PWB, SWB, EWB, FWB, and LeuS, respectively. FACT-Leu total score ranged from 0 to 176. Higher scores indicated a better quality of life. Best change from baseline was defined as the highest value of change from baseline among all postbaseline visits. For participants who did not enter Study GS-US-312-0117, baseline values were from Study GS-US-312-0116.
Time Frame: Study GS-US-312-0116 or GS-US-312-0117 Baseline up to Week 184
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IDL+R to IDL | Placebo+R (PD) to IDL 150 mg | Placebo+R to IDL 150 mg
Number analyzed (Participants) | 107 | 42 | 44
units on a scale
  Total Score: Baseline: number analyzed (Participants) | 103 | 42 | 43
  Total Score: Baseline | 128.4 (22.72) | 116.7 (29.56) | 128.1 (29.16)
  PWB: Baseline: number analyzed (Participants) | 106 | 42 | 44
  PWB: Baseline | 22.8 (4.42) | 20.2 (5.93) | 21.9 (5.41)
  SWB: Baseline: number analyzed (Participants) | 107 | 42 | 43
  SWB: Baseline | 22.5 (5.53) | 22.5 (5.06) | 23.5 (5.04)
  EWB: Baseline: number analyzed (Participants) | 104 | 42 | 44
  EWB: Baseline | 19.1 (3.44) | 17.3 (4.97) | 17.6 (4.48)
  FWB: Baseline: number analyzed (Participants) | 106 | 42 | 44
  FWB: Baseline | 18.0 (6.57) | 15.0 (7.17) | 18.0 (6.88)
  LeuS: Baseline: number analyzed (Participants) | 106 | 42 | 44
  LeuS: Baseline | 46.0 (10.64) | 41.7 (12.74) | 47.0 (12.01)
  Total Score: Best Change from Baseline: number analyzed (Participants) | 101 | 39 | 40
  Total Score: Best Change from Baseline | 21.8 (19.64) | 20.2 (19.91) | 14.9 (12.04)
  PWB: Best Change from Baseline: number analyzed (Participants) | 102 | 39 | 40
  PWB: Best Change from Baseline | 3.1 (4.65) | 3.6 (4.26) | 3.4 (3.81)
  SWB: Best Change from Baseline: number analyzed (Participants) | 104 | 39 | 39
  SWB: Best Change from Baseline | 2.9 (5.21) | 2.0 (2.88) | 2.1 (2.39)
  EWB: Best Change from Baseline: number analyzed (Participants) | 101 | 39 | 40
  EWB: Best Change from Baseline | 3.1 (2.75) | 3.1 (3.68) | 2.8 (3.14)
  FWB: Best Change from Baseline: number analyzed (Participants) | 104 | 39 | 38
  FWB: Best Change from Baseline | 5.1 (5.80) | 4.1 (5.01) | 3.1 (2.94)
  LeuS: Best Change from Baseline: number analyzed (Participants) | 104 | 39 | 41
  LeuS: Best Change from Baseline | 11.3 (9.13) | 10.1 (8.78) | 7.8 (5.59)

17. Secondary Outcome: Best Change From Baseline in Karnofsky Performance Status (KPS)
Description: KPS is a tool used to measure the ability to perform ordinary tasks. The score ranges from 0 to 100, with a higher score indicating that the participant is better able to carry out daily activities. Best change from baseline was defined as the highest value of change from baseline among all postbaseline visits. For participants who did not enter Study GS-US-312-0117, baseline values were from Study GS-US-312-0116.
Time Frame: Study GS-US-312-0116 or GS-US-312-0117 Baseline up to Week 190
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IDL+R to IDL | Placebo+R (PD) to IDL 150 mg | Placebo+R to IDL 150 mg
Number analyzed (Participants) | 110 | 42 | 44
units on a scale
  Baseline | 80.7 (12.47) | 78.1 (14.18) | 86.8 (8.83)
  Best Change From Baseline: number analyzed (Participants) | 105 | 38 | 35
  Best Change From Baseline | 11.1 (10.31) | 7.1 (8.67) | 4.3 (6.98)

18. Secondary Outcome: Changes From Baseline in Phosphatidylinositol 3-kinase (PI3Kδ)/Akt/Mammalian Target of Rapamycin (mTOR) Pathway Activation as a Measure of PI3Kδ Pathway Activity
Time Frame: GS-US-312-0116 Baseline to end of study GS-US-312-0117 (maximum: up to 67.6 months)
Population: Data were not collected because there was insufficient volume of sample (not enough material) to perform the analysis for any participant.
Groups:
- IDL+R to IDL: Participants received IDL 150 mg tablet twice daily plus rituximab (8 infusions intravenously) in Study GS-US-312-0116 and may have entered Study GS-US-312-0117 to receive IDL 150 mg or 300 mg tablet twice daily.
Arm/Group | IDL+R to IDL | Placebo+R (PD) to IDL 150 mg | Placebo+R to IDL 150 mg
Number analyzed (Participants) | 0 | 0 | 0

19. Secondary Outcome: Overall Change From Baseline in the Plasma Concentrations of Disease-Associated Chemokines and Cytokines
Description: The percent of average on-treatment biomarker concentration of baseline (%Baseline) was used to evaluate the overall pharmacodynamics change on the biomarkers with IDL treatment. The average on-treatment biomarker concentration is calculated using area under curve (AUC) following the trapezoidal rule. The biomarkers with median AUC value of 100 indicated no overall on-treatment biomarker changes compared to the baseline. The biomarkers with median AUC value greater than 100 or less than 100 indicated an increase or decrease, respectively, on-treatment biomarker changes from the baseline.
Time Frame: GS-US-312-0116 Baseline to end of study GS-US-312-0117 (maximum: up to 67.6 months)
Population: The cytokine and T-cell subsets biomarker analysis set included all participants who received at least one dose of study drug, consented for optional future study, and had at least one evaluable measurement for any biomarker at any visit on IDL treatment. Available samples were batched for analysis as prespecified.
Measure: Median (Full Range); unit: percentage of baseline
Groups:
- IDL/Placebo+R to IDL: Participants received IDL 150 mg tablet or placebo tablet twice daily plus rituximab (8 infusions intravenously) in Study GS-US-312-0116 (either met or not met the primary endpoint of PD) and may have entered Study GS-US-312-0117 to receive IDL 150 mg or 300 mg tablet twice daily.
Arm/Group | IDL/Placebo+R to IDL
Number analyzed (Participants) | 174
percentage of baseline
  Tumor Necrosis Factor (TNF)-alpha | 36.73 [5.34 to 183.56]
  Macrophage Inflammatory Protein (MIP)1-alpha | 26.55 [3.76 to 236.22]
  Interleukin (IL)-10 | 58.65 [2.36 to 1706.34]
  IL-15 | 111.18 [51.28 to 230.1]
  IL-12p40 | 64.89 [11.3 to 2012.31]
  RANTES (CCL5) | 131.94 [6.76 to 3715.99]
  IL-1ra | 114.22 [11.64 to 608.17]
  Interferon (IFN)-gamma | 127.72 [10.55 to 4736.96]
  C-Reactive Protein (CRP) | 132.38 [9.67 to 7625.53]
  IFN-gamma-induced protein (IP)-10 (CXCL10) | 88.5 [15.24 to 786.21]
  IL-7 | 91.82 [14.47 to 960.7]
  Granulocyte-colony stimulating factor (G-CSF) | 96.59 [3.83 to 1586.48]
  IL-17A | 100 [8.8 to 1311.69]
  IL-6 | 100 [7.13 to 2817.44]
  IL-8 | 102.59 [2.47 to 1724.25]

20. Secondary Outcome: Study Drug Compliance as Assessed by the Percentage of Participants Adhering to Treatment
Description: Adherence percentage was calculated as the sum of tablets dispensed - the sum of tablets returned divided by the sum of the overall dosing period (total daily tablets x dosing duration), taking into account investigator-prescribed interruptions.
Time Frame: First IDL dose date in study GS-US-312-0116 or GS-US-312-0117 to last IDL dose date in study GS-US-312-0117 (maximum: 67.3 months)
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | IDL+R to IDL | Placebo+R (PD) to IDL 150 mg | Placebo+R to IDL 150 mg
Number analyzed (Participants) | 110 | 42 | 44
percentage of participants
  Adherence ≥ 75% | 100.0 | 97.6 | 100.0
  Adherence < 75% | 0.0 | 2.4 | 0.0

21. Secondary Outcome: Plasma Trough (Predose) and Peak (1.5 Hours Postdose) Concentrations of Idelalisib
Time Frame: Weeks 4, 12, and 24
Population: Participants in the pharmacokinetic (PK) Analysis Set (participants in the Full Analysis Set who had the necessary baseline and on-study measurements to provide interpretable results for the specific parameters of interest) with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Groups:
- IDL+R to IDL 150 mg: Participants who received IDL 150 mg tablet twice daily plus rituximab (8 infusions intravenously) in Study GS-US-312-0116 and entered Study GS-US-312-0117 to receive IDL 150 mg tablet twice daily.
- IDL+R (PD) to IDL 300 mg: Participants received IDL 150 mg tablet twice daily plus rituximab (8 infusions intravenously) in Study GS-US-312-0116 and met the primary endpoint of PD and entered Study GS-US-312-0117 to receive IDL 300 mg tablet twice daily.
Arm/Group | IDL+R to IDL 150 mg | IDL+R (PD) to IDL 300 mg | Placebo+R (PD) to IDL 150 mg | Placebo+R to IDL 150 mg
Number analyzed (Participants) | 40 | 3 | 30 | 29
ng/mL
  Week 4: Predose | 384.0 [166.5 to 681.5] | 470.0 [317.0 to 631.0] | 301.5 [195.0 to 494.0] | 412.0 [211.0 to 646.0]
  Week 4: 1.5 Hours Postdose: number analyzed (Participants) | 38 | 3 | 29 | 29
  Week 4: 1.5 Hours Postdose | 2115.0 [1370.0 to 2750.0] | 3940.0 [1550.0 to 4000.0] | 2580.0 [1880.0 to 3080.0] | 1720.0 [1200.0 to 2660.0]
  Week 12: Predose: number analyzed (Participants) | 35 | 3 | 29 | 26
  Week 12: Predose | 370.0 [196.0 to 745.0] | 570.0 [355.0 to 643.0] | 335.0 [190.0 to 470.0] | 298.0 [212.0 to 691.0]
  Week 12: 1.5 Hours Postdose: number analyzed (Participants) | 32 | 3 | 28 | 26
  Week 12: 1.5 Hours Postdose | 2110.0 [1595.0 to 2665.0] | 3800.0 [3160.0 to 4710.0] | 2245.0 [1655.0 to 3255.0] | 1940.0 [1430.0 to 2450.0]
  Week 24: Predose: number analyzed (Participants) | 33 | 3 | 19 | 16
  Week 24: Predose | 307.0 [179.0 to 584.0] | 637.0 [524.0 to 930.0] | 362.0 [162.0 to 550.0] | 350.5 [261.0 to 504.5]
  Week 24: 1.5 Hours Postdose: number analyzed (Participants) | 34 | 3 | 19 | 17
  Week 24: 1.5 Hours Postdose | 2270.0 [1560.0 to 2790.0] | 5630.0 [5550.0 to 5660.0] | 2180.0 [1760.0 to 2980.0] | 2010.0 [1210.0 to 2430.0]

22. Secondary Outcome: Change in Health Status as Assessed Using the EuroQoL Five-Dimension (EQ-5D) Utility Measure
Description: Change in health status was defined as the change from baseline in overall health and single-item dimension scores as assessed using the EQ-5D utility measure. Percentage of participants with different level of problem were reported. Level 1: indicated no problem; Level 2: indicated some problems; and Level 3: indicated extreme problems. For participants who did not enter Study GS-US-312-0117, baseline values were from Study GS-US-312-0116.
Time Frame: Study GS-US-312-0116 or GS-US-312-0117 Baseline; Weeks 24 and 48
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | IDL+R to IDL | Placebo+R (PD) to IDL 150 mg | Placebo+R to IDL 150 mg
Number analyzed (Participants) | 108 | 42 | 44
percentage of participants
  Baseline: Anxiety/Depression, Level 1 | 70.4 | 50.0 | 56.8
  Baseline: Anxiety/Depression, Level 2 | 28.7 | 42.9 | 43.2
  Baseline: Anxiety/Depression, Level 3 | 0.9 | 7.1 | 0.0
  Baseline: Mobility, Level 1 | 60.2 | 38.1 | 61.4
  Baseline: Mobility, Level 2 | 39.8 | 59.5 | 38.6
  Baseline: Mobility, Level 3 | 0.0 | 2.4 | 0.0
  Baseline: Pain/Discomfort, Level 1 | 53.3 | 50.0 | 45.5
  Baseline: Pain/Discomfort, Level 2 | 39.3 | 45.2 | 50.0
  Baseline: Pain/Discomfort, Level 3 | 7.5 | 4.8 | 4.5
  Baseline: Self-Care, Level 1 | 90.7 | 76.2 | 84.1
  Baseline: Self-Care, Level 2 | 9.3 | 19.0 | 15.9
  Baseline: Self-Care, Level 3 | 0.0 | 4.8 | 0.0
  Baseline: Usual Activities, Level 1 | 56.5 | 28.6 | 52.3
  Baseline: Usual Activities, Level 2 | 36.1 | 52.4 | 45.5
  Baseline: Usual Activities, Level 3 | 7.4 | 19.0 | 2.3
  Week 24: Anxiety/Depression, Level 1: number analyzed (Participants) | 77 | 20 | 23
  Week 24: Anxiety/Depression, Level 1 | 83.1 | 65.0 | 69.6
  Week 24: Anxiety/Depression, Level 2: number analyzed (Participants) | 77 | 20 | 23
  Week 24: Anxiety/Depression, Level 2 | 15.6 | 35.0 | 30.4
  Week 24: Anxiety/Depression, Level 3: number analyzed (Participants) | 77 | 20 | 23
  Week 24: Anxiety/Depression, Level 3 | 1.3 | 0.0 | 0.0
  Week 24: Mobility, Level 1: number analyzed (Participants) | 77 | 20 | 23
  Week 24: Mobility, Level 1 | 70.1 | 65.0 | 69.6
  Week 24: Mobility, Level 2: number analyzed (Participants) | 77 | 20 | 23
  Week 24: Mobility, Level 2 | 29.9 | 35.0 | 30.4
  Week 24: Mobility, Level 3: number analyzed (Participants) | 77 | 20 | 23
  Week 24: Mobility, Level 3 | 0.0 | 0.0 | 0.0
  Week 24: Pain/Discomfort, Level 1: number analyzed (Participants) | 77 | 20 | 23
  Week 24: Pain/Discomfort, Level 1 | 62.3 | 65.0 | 43.5
  Week 24: Pain/Discomfort, Level 2: number analyzed (Participants) | 77 | 20 | 23
  Week 24: Pain/Discomfort, Level 2 | 35.1 | 30.0 | 47.8
  Week 24: Pain/Discomfort, Level 3: number analyzed (Participants) | 77 | 20 | 23
  Week 24: Pain/Discomfort, Level 3 | 2.6 | 5.0 | 8.7
  Week 24: Self-Care, Level 1: number analyzed (Participants) | 77 | 20 | 23
  Week 24: Self-Care, Level 1 | 92.2 | 85.0 | 91.3
  Week 24: Self-Care, Level 2: number analyzed (Participants) | 77 | 20 | 23
  Week 24: Self-Care, Level 2 | 6.5 | 15.0 | 8.7
  Week 24: Self-Care, Level 3: number analyzed (Participants) | 77 | 20 | 23
  Week 24: Self-Care, Level 3 | 1.3 | 0.0 | 0.0
  Week 24: Usual Activities, Level 1: number analyzed (Participants) | 77 | 20 | 23
  Week 24: Usual Activities, Level 1 | 68.4 | 75.0 | 60.9
  Week 24: Usual Activities, Level 2: number analyzed (Participants) | 77 | 20 | 23
  Week 24: Usual Activities, Level 2 | 28.9 | 25.0 | 34.8
  Week 24: Usual Activities, Level 3: number analyzed (Participants) | 77 | 20 | 23
  Week 24: Usual Activities, Level 3 | 2.6 | 0.0 | 4.3
  Week 48: Anxiety/Depression, Level 1: number analyzed (Participants) | 44 | 10 | 6
  Week 48: Anxiety/Depression, Level 1 | 84.1 | 90.0 | 50.0
  Week 48: Anxiety/Depression, Level 2: number analyzed (Participants) | 44 | 10 | 6
  Week 48: Anxiety/Depression, Level 2 | 15.9 | 10.0 | 50.0
  Week 48: Anxiety/Depression, Level 3: number analyzed (Participants) | 44 | 10 | 6
  Week 48: Anxiety/Depression, Level 3 | 0.0 | 0.0 | 0.0
  Week 48: Mobility, Level 1: number analyzed (Participants) | 44 | 10 | 6
  Week 48: Mobility, Level 1 | 72.7 | 60.0 | 66.7
  Week 48: Mobility, Level 2: number analyzed (Participants) | 44 | 10 | 6
  Week 48: Mobility, Level 2 | 27.3 | 40.0 | 33.3
  Week 48: Mobility, Level 3: number analyzed (Participants) | 44 | 10 | 6
  Week 48: Mobility, Level 3 | 0.0 | 0.0 | 0.0
  Week 48: Pain/Discomfort, Level 1: number analyzed (Participants) | 44 | 10 | 6
  Week 48: Pain/Discomfort, Level 1 | 56.8 | 60.0 | 50.0
  Week 48: Pain/Discomfort, Level 2: number analyzed (Participants) | 44 | 10 | 6
  Week 48: Pain/Discomfort, Level 2 | 43.2 | 30.0 | 50.0
  Week 48: Pain/Discomfort, Level 3: number analyzed (Participants) | 44 | 10 | 6
  Week 48: Pain/Discomfort, Level 3 | 0.0 | 10.0 | 0.0
  Week 48: Self-Care, Level 1: number analyzed (Participants) | 44 | 10 | 6
  Week 48: Self-Care, Level 1 | 95.5 | 90.0 | 83.3
  Week 48: Self-Care, Level 2: number analyzed (Participants) | 44 | 10 | 6
  Week 48: Self-Care, Level 2 | 4.5 | 0.0 | 16.7
  Week 48: Self-Care, Level 3: number analyzed (Participants) | 44 | 10 | 6
  Week 48: Self-Care, Level 3 | 0.0 | 10.0 | 0.0
  Week 48: Usual Activities, Level 1: number analyzed (Participants) | 44 | 10 | 6
  Week 48: Usual Activities, Level 1 | 72.7 | 70.0 | 50.0
  Week 48: Usual Activities, Level 2: number analyzed (Participants) | 44 | 10 | 6
  Week 48: Usual Activities, Level 2 | 25.0 | 20.0 | 33.3
  Week 48: Usual Activities, Level 3: number analyzed (Participants) | 44 | 10 | 6
  Week 48: Usual Activities, Level 3 | 2.3 | 10.0 | 16.7

ADVERSE EVENTS:
Time Frame: Adverse Events: First IDL dose date in study GS-US-312-0116 or GS-US-312-0117 to last IDL dose date in study GS-US-312-0117 (maximum: 67.3 months) plus 30 days; All-Cause Mortality: First IDL dose date up to 67.6 months
Description: Only adverse events occurring in participants who enrolled into the extension Study GS-US-312-0117 were included. Adverse events occurring in the parent study, GS-US-312-0116, are reported in ClinicalTrials.gov record NCT01539512.
Groups:
- IDL+R to IDL 150 mg: Adverse events reported in this group occurred during the extension Study GS-US-312-0117 in participants who received IDL 150 mg tablet twice daily plus rituximab (8 infusions intravenously) in Study GS-US-312-0116 and entered Study GS-US-312-0117 to receive IDL 150 mg tablet twice daily.
- IDL+R (PD) to IDL 300 mg: Adverse events reported in this group occurred during the extension Study GS-US-312-0117 in participants who received IDL 150 mg tablet twice daily plus rituximab (8 infusions intravenously) in Study GS-US-312-0116 and entered Study GS-US-312-0117 to receive IDL 300 mg tablet twice daily.
- Placebo+R (PD) to IDL 150 mg: Adverse events reported in this group occurred during the extension Study GS-US-312-0117 in participants who received placebo tablet twice daily plus rituximab (8 infusions intravenously) in Study GS-US-312-0116 and met the primary endpoint of PD and entered Study GS-US-312-0117 to receive IDL 150 mg tablet twice daily.
- Placebo+R to IDL 150 mg: Adverse events reported in this group occurred during the extension Study GS-US-312-0117 in participants who received placebo tablet twice daily plus rituximab (8 infusions intravenously) in Study GS-US-312-0116 and entered Study GS-US-312-0117 to receive IDL 150 mg tablet twice daily.
Arm/Group | IDL+R to IDL 150 mg | IDL+R (PD) to IDL 300 mg | Placebo+R (PD) to IDL 150 mg | Placebo+R to IDL 150 mg
All-Cause Mortality (participants affected / at risk) | 37/71 | 3/4 | 25/42 | 16/44
Serious Adverse Events (participants affected / at risk) | 54/71 | 2/4 | 34/42 | 32/44
Other Adverse Events (participants affected / at risk) | 70/71 | 4/4 | 41/42 | 43/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IDL+R to IDL 150 mg (N=71) | IDL+R (PD) to IDL 300 mg (N=4) | Placebo+R (PD) to IDL 150 mg (N=42) | Placebo+R to IDL 150 mg (N=44)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 0 | 5 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 2
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 2 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 5 | 0 | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 7 | 0 | 4 | 8
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 2 | 1
Drug withdrawal syndrome (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 2
General physical health deterioration (General disorders) | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 4 | 0 | 1 | 4
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 1
Acute sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 1
Candida infection (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 4 | 0 | 0 | 4
Cerebral fungal infection (Infections and infestations) | 0 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1 | 0
Encephalitis (Infections and infestations) | 0 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 5 | 0 | 0 | 3
Lung infection (Infections and infestations) | 1 | 0 | 0 | 0
Mastoiditis (Infections and infestations) | 0 | 0 | 1 | 0
Neutropenic sepsis (Infections and infestations) | 2 | 0 | 1 | 0
Oesophageal infection (Infections and infestations) | 0 | 0 | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 6 | 2 | 10 | 3
Pneumonia escherichia (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia haemophilus (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia influenzal (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia pseudomonal (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia viral (Infections and infestations) | 1 | 0 | 0 | 0
Progressive multifocal leukoencephalopathy (Infections and infestations) | 1 | 0 | 0 | 0
Pseudomonal bacteraemia (Infections and infestations) | 0 | 0 | 1 | 1
Pseudomonal sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Pseudomonas infection (Infections and infestations) | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 5 | 0 | 1 | 0
Sepsis pasteurella (Infections and infestations) | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 2 | 0 | 1 | 2
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis fungal (Infections and infestations) | 0 | 0 | 0 | 1
Stenotrophomonas infection (Infections and infestations) | 0 | 0 | 1 | 0
Streptococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 1
Tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Feeding intolerance (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Lung squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Melanoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 1
Central nervous system haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1 | 0 | 0
Aortic dissection (Vascular disorders) | 1 | 0 | 0 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 0 | 0 | 1
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Shock haemorrhagic (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IDL+R to IDL 150 mg (N=71) | IDL+R (PD) to IDL 300 mg (N=4) | Placebo+R (PD) to IDL 150 mg (N=42) | Placebo+R to IDL 150 mg (N=44)
Anaemia (Blood and lymphatic system disorders) | 8 | 2 | 5 | 4
Neutropenia (Blood and lymphatic system disorders) | 14 | 1 | 9 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 2 | 3 | 4
Abdominal distension (Gastrointestinal disorders) | 3 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 8 | 1 | 5 | 5
Colitis (Gastrointestinal disorders) | 1 | 0 | 4 | 6
Constipation (Gastrointestinal disorders) | 11 | 1 | 7 | 4
Diarrhoea (Gastrointestinal disorders) | 30 | 2 | 17 | 26
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 4 | 0 | 2 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Flatulence (Gastrointestinal disorders) | 2 | 0 | 0 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 1 | 5 | 2
Haemorrhoids (Gastrointestinal disorders) | 2 | 0 | 4 | 6
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 2 | 0
Nausea (Gastrointestinal disorders) | 11 | 0 | 12 | 12
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 3
Vomiting (Gastrointestinal disorders) | 7 | 0 | 7 | 9
Asthenia (General disorders) | 5 | 0 | 7 | 2
Chills (General disorders) | 7 | 0 | 6 | 4
Fatigue (General disorders) | 15 | 2 | 13 | 9
Malaise (General disorders) | 2 | 0 | 2 | 3
Mucosal inflammation (General disorders) | 1 | 0 | 1 | 3
Oedema (General disorders) | 0 | 0 | 0 | 3
Oedema peripheral (General disorders) | 12 | 0 | 7 | 8
Pain (General disorders) | 3 | 0 | 3 | 5
Peripheral swelling (General disorders) | 1 | 0 | 1 | 3
Pyrexia (General disorders) | 17 | 0 | 12 | 16
Hypogammaglobulinaemia (Immune system disorders) | 3 | 0 | 2 | 4
Bronchitis (Infections and infestations) | 4 | 1 | 2 | 6
Cellulitis (Infections and infestations) | 4 | 0 | 0 | 2
Ear infection (Infections and infestations) | 4 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 2 | 0 | 2 | 3
Lower respiratory tract infection (Infections and infestations) | 3 | 0 | 1 | 4
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 5
Oral candidiasis (Infections and infestations) | 2 | 0 | 0 | 3
Pharyngitis (Infections and infestations) | 1 | 0 | 1 | 4
Pneumonia (Infections and infestations) | 4 | 0 | 9 | 6
Sinusitis (Infections and infestations) | 14 | 1 | 1 | 4
Upper respiratory tract infection (Infections and infestations) | 10 | 0 | 8 | 11
Urinary tract infection (Infections and infestations) | 7 | 0 | 3 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 3 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 3
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 3 | 1 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 3
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 3
Computerised tomogram thorax abnormal (Investigations) | 1 | 1 | 0 | 1
Weight decreased (Investigations) | 5 | 1 | 4 | 5
Decreased appetite (Metabolism and nutrition disorders) | 9 | 1 | 1 | 6
Dehydration (Metabolism and nutrition disorders) | 6 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 4 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 0 | 3 | 7
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 0 | 3 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 0 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 1 | 5 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 0 | 2 | 3
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 0 | 5 | 5
Headache (Nervous system disorders) | 6 | 0 | 3 | 6
Lethargy (Nervous system disorders) | 6 | 0 | 3 | 1
Device occlusion (Product Issues) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 0 | 3 | 2
Depression (Psychiatric disorders) | 3 | 0 | 0 | 3
Insomnia (Psychiatric disorders) | 6 | 0 | 3 | 2
Acute kidney injury (Renal and urinary disorders) | 6 | 0 | 1 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 3
Haematuria (Renal and urinary disorders) | 5 | 1 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 4 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 21 | 0 | 12 | 16
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 0 | 4 | 10
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 3 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 1 | 0
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 4 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 7 | 0 | 0 | 7
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 4 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 3
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 3
Night sweats (Skin and subcutaneous tissue disorders) | 6 | 1 | 10 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 3
Rash (Skin and subcutaneous tissue disorders) | 5 | 0 | 4 | 7
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 0 | 2 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 3 | 0 | 2 | 3
Hypertension (Vascular disorders) | 4 | 0 | 0 | 2
Hypotension (Vascular disorders) | 4 | 0 | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (12):
  • Study Protocol: Original (2012-01-23): https://cdn.clinicaltrials.gov/large-docs/91/NCT01539291/Prot_000.pdf
  • Study Protocol: Amendment 1 (2013-01-23): https://cdn.clinicaltrials.gov/large-docs/91/NCT01539291/Prot_001.pdf
  • Study Protocol: Amendment 2 (2013-09-10): https://cdn.clinicaltrials.gov/large-docs/91/NCT01539291/Prot_002.pdf
  • Study Protocol: Amendment 3 (2013-12-16): https://cdn.clinicaltrials.gov/large-docs/91/NCT01539291/Prot_003.pdf
  • Study Protocol: Amendment 4 (2014-05-27): https://cdn.clinicaltrials.gov/large-docs/91/NCT01539291/Prot_004.pdf
  • Study Protocol: Amendment 5 (2014-10-10): https://cdn.clinicaltrials.gov/large-docs/91/NCT01539291/Prot_005.pdf
  • Study Protocol: Amendment 6 (2016-03-28): https://cdn.clinicaltrials.gov/large-docs/91/NCT01539291/Prot_006.pdf
  • Study Protocol: Amendment 7 (2016-08-05): https://cdn.clinicaltrials.gov/large-docs/91/NCT01539291/Prot_007.pdf
  • Statistical Analysis Plan: Blinded (2013-11-04): https://cdn.clinicaltrials.gov/large-docs/91/NCT01539291/SAP_008.pdf
  • Statistical Analysis Plan: Open Label (2015-01-26): https://cdn.clinicaltrials.gov/large-docs/91/NCT01539291/SAP_009.pdf
  • Study Protocol: Amendment 8 (2016-10-24): https://cdn.clinicaltrials.gov/large-docs/91/NCT01539291/Prot_010.pdf
  • Study Protocol: Amendment 9 (2017-09-21): https://cdn.clinicaltrials.gov/large-docs/91/NCT01539291/Prot_011.pdf